CLINICAL TRIAL: NCT00867737
Title: Onset of Action of Advair HFA 115/21 in Comparison to Symbicort pMDI 160/4.5 Measured by Impulse Oscillometry, IOS.
Brief Title: Onset of Action of Advair Hydrofluoroalkane (HFA) 115/21 in Comparison to Symbicort Pressurised Metered-Dose Inhalers (pMDI) 160/4.5 Measured by Impulse Oscillometry (IOS)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Allergy and Asthma Center of El Paso (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Rogelio Menendez, MD/Principal Investigator, Allergy and Asthma Center of El Paso
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRT112430
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Last update posted 2009-03-24 (Estimated); Status verified 2009-03

CONDITIONS: Asthma
Keywords: Asthma; Forced Oscillation; Impulse Oscillometry; Electrical-equivalent respiratory system model
MeSH Terms: conditions — Asthma | interventions — Salmeterol Xinafoate; Formoterol Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Advair 115/21 MDI (Experimental): Advair HFA 115/21 MDI Intervention = initiate intervention after screening
  Interventions: Drug: Advair HFA MDI 115/21
- 2 = Symbicort 160/4.5 (Active Comparator): Symbicort initiated after screening
  Interventions: Drug: Symbicort 160/4.5 pMDI

INTERVENTIONS:
Drug: Advair HFA MDI 115/21 — Two puffs from MDI twice daily for 4 weeks
  Other Names: Advair = fluticasone proprionate plus salmeterol
  Arms: Advair 115/21 MDI
Drug: Symbicort 160/4.5 pMDI — Symbicort 160/4.5 pMDI
  Two puffs from MDI twice daily for 4 weeks
  Other Names: Symbicort = budesonide plus formoterol fumarate
  Arms: 2 = Symbicort 160/4.5

SUMMARY:
The objectives of this study are to measure Impulse Oscillometry (IOS) in patients with asthma extensively at baseline in patients with mild-to-moderate asthma, treated with as-needed short acting beta agonist only, to measure respiratory resistance and small airway dysfunction accurately and precisely at baseline, from which to measure onset of action of Advair MDI in comparison with that of Symbicort MDI. Initial screening will assess IOS resistance and small airway dysfunction and its response to short acting beta agonist (SABA). Patients will be selected from among those who manifest a 40% improvement in small airway function assessed by IOS low frequency reactance after SABA compared to baseline. After screening, patients will be randomized to receive either Advair or Symbicort; and will be assessed at randomization before and at several intervals after initial dosing, up to 4 hours. Patients will return again 4 weeks after randomization for extended IOS (and spirometry) testing as done at randomization.

DETAILED DESCRIPTION:
Eligibility criteria include age 12-45 years, with current treatment of asthma with as-needed SABA only; and manifesting an acute response to SABA at screening of 40% or greater improvement in IOS low frequency reactance. After inclusion in the protocol, all subjects will receive active treatment, either with Advair or with Symbicort. Outcome measures will include large and small airway resistance and integrated low-frequency reactance calculated directly from IOS measures, and in addition, Large Airway Resistance, Small Airway Resistance and Small Airway Compliance derived from an electrical equivalent respiratory system model. Analysis of IOS data will be done post-testing by a respiratory physiologist, experienced with use of IOS and its analysis and interpretation, blinded to which treatment each individual received. Electrical-equivalent respiratory system model analyses will be done by a biomedical engineer, blinded to which treatment each individual received.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of asthma
* Asthma symptoms controlled by short-acting beta agonist as-needed
* Age 12-45 years

Exclusion Criteria:

* Severe asthma
* use of oral or inhaled corticosteroids within 30 days of screening

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-09 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Integrated low frequency reactance improvement after initial dosing | 5, 20, 40, 60, 120, and 240 min

SECONDARY OUTCOMES:
Frequency-dependence of Resistance (R5-R20) after initial dosing | 5, 20, 40, 60, 120, and 240 min
Model-derived estimates of Large and Small Airway Resistance and Compliance, and their changes after initial dosing | 5, 20, 40, 60, 120, and 240 min

CONTACTS AND LOCATIONS:
Overall Officials: Rogelio Menendez, MD, Principal Investigator — Allergy and Asthma Center of El Paso
Locations (1):
- Allergy and Asthma Center of El Paso, El Paso, Texas, United States